CLINICAL TRIAL: NCT00649168
Title: Study of Mylan Pharmaceuticals Inc. and Novartis Pharmaceuticals Corporation (Parlodel®) 5 mg Bromocriptine Mesylate Capsules Following a 10 mg Dose in Healthy Adult Volunteers Under Fed Conditions
Brief Title: Fed Study of (Parlodel®) Bromocriptine Mesylate Capsules 5 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BROM-0733
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Bromocriptine; Capsules

ARMS (2):
- 1 (Experimental): Metoclopramide Hydrochloride Injection Sandoz Standard 5mg/mL (10mg/2mL)and BROMOCRIPTINE MESYLATE CAPSULES, USP 5 mg
  Interventions: Drug: BROMOCRIPTINE MESYLATE CAPSULES, USP 5 mg
- 2 (Active Comparator): Metoclopramide Hydrochloride Injection Sandoz Standard 5mg/mL (10mg/2mL) and Parlodel® (bromocriptine mesylate) capsules, USP 5 mg
  Interventions: Drug: Parlodel® (bromocriptine mesylate) capsules, USP 5 mg

INTERVENTIONS:
Drug: BROMOCRIPTINE MESYLATE CAPSULES, USP 5 mg — 2x5mg bromocriptine mesylate, single dose fed; with 10mg metoclopramide HCl prophylactic injection
  Arms: 1
Drug: Parlodel® (bromocriptine mesylate) capsules, USP 5 mg — 2x5mg bromocriptine mesylate, single dose fed; with 10mg metoclopramide HCl prophylactic injection
  Arms: 2

SUMMARY:
The objective of this study was to assess the single-dose relative bioavailability of Mylan Pharmaceuticals Inc. and Novartis Pharmaceuticals Corporation (Parlodel®) 5 mg bromocriptine mesylate capsules, following the administration of a 10 mg dose, under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult male or female volunteers, 18-45 years of age Subjects will be continuous non-smokers for at least 3 months prior to the first dose or consistent moderate smokers (fewer than 10 cigarettes per day) for at least 3 months prior to the first dosing Weighing at least 60 kg for males and 52 kg for females and within the normal range, according to accepted normal values of the Body Mass Index chart (BMI) (18.00-28.00 kg/m2) Medically healthy subjects with clinically normal laboratory profiles and 12-lead ECG Females of childbearing potential should either be sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or be using one of the following acceptable birth control methods surgically sterile (bilateral tubal ligation hysterectomy bilateral oophorectomy) 6 months minimum IUD (excluding hormone-releasing-IUD) in place for at least 3 months and throughout the study barrier methods (condom or diaphragm) with spermicide for at least 14 days prior to the first dose and throughout the study surgical sterilization of the partner (vasectomy for 6 months minimum) In addition female subjects of childbearing potential will be advised to remain sexually inactive or to keep the same birth control method for at least 3 days following the last dose Other birth control methods may be deemed acceptable Postmenopausal women with amenorrhea for at least 2 years will be eligible. Males must use a spermicide-containing barrier method of contraception to prevent the pregnancy of their female sexual partner from screening, throughout the entire study and for at least 3 days following the last dose Give voluntary written informed consent to participate in the study

Exclusion Criteria:

History or presence of significant cardiovascular pulmonary hepatic renal, hematologic gastrointestinal endocrine immunologic dermatologic neurologic or psychiatric disease In addition history or presence of depression seizure or history of EEG abnormalities glaucoma or hypermetropia frequent migraine episodes alcoholism or drug abuse within the past year past psychotic or maniac episodes asthma chronic bronchitis or any other bronchospastic conditions peptic ulcer hypersensitivity or idiosyncratic reaction to bromocriptine or to any ergot alkaloids related compound hypersensitivity or idiosyncratic reaction to acetaminophen diphenhydramine metoclopramide diazepam or any phenothiazines related compound subjects who tested positive at screening for HIV, HbsAg or HCV Subjects whose sitting blood pressure is less than 110/60 mmHg at screening or less than 100/55 mmHg prior to dosing in each period Subjects whose sitting blood pressure is more than 140/90 mmHg at screening or prior to dosing in each period Subjects whose pulse is lower than 55 b.p.m. at screening or 50 b.p.m. prior to dosing in each period Female subjects who are pregnant or lactating Female subjects who are taking hormonal contraceptives or are on hormonal replacement therapy (this includes all formulation, e.g. oral, transdermal, vaginal) during the 28 days prior to the first dose and throughout the study Subjects who have used Depo-Provera® or levonorgestrel implant within 90 days prior to the first dose and throughout the study Subjects who have received any substance with monoamine oxidase inhibitor (MAOI) activity within 28 days prior to the first dose Subjects who have food allergy, problems of galactose intolerance or glucose-galactose malabsorption, or any restriction that, in the opinion of the Principal Investigator, could contraindicate the subject's participation in the study Subjects who have been on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study Subjects who donated 50 to 499 mL of blood within 30 days and more than 499 mL within 56 days prior to the first dose Subjects who, through completion of the study would have donated in excess of 500 mL of blood in 14 days 1500 mL of blood in 180 days 2500 mL of blood in 1 year Subjects who have participated in another clinical trial within 28 days prior to the first dose

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2007-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli, M.D., Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Montreal, Quebec, Canada

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html